CLINICAL TRIAL: NCT01729377
Title: The Meaning of Suicidality for Older Persons With Suicidal Tendencies and Their Families
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: 290466-HYMC
Record Dates: First submitted 2012-11-14; First posted 2012-11-20 (Estimated); Last update posted 2012-11-20 (Estimated); Status verified 2012-11

CONDITIONS: Suicide; Aged; Family
MeSH Terms: conditions — Suicide | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Suicidal older persons and their families: Suicidal older persons and their families will be interviewed
  Interventions: Other: Interview

INTERVENTIONS:
Other: Interview

SUMMARY:
The purpose of the proposed study is to examine the phenomenon of suicidality in old age and its unique characteristics. This will be performed through observing the multigenerational aging family from the life-course perspective, which enables the researchers to address life transitions, including crises leading to suicidal tendencies.

ELIGIBILITY:
Inclusion Criteria:

* Hebrew speaking
* Suicidal
* Families of elderly suicides
* Cognitive ability

Exclusion Criteria:

* All others

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Aged individuals from tertiary and primary care and from the community who have experienced suicidality and their families.
Sampling Method: Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2013-04; Primary Completion 2014-04 (Estimated); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
Understanding older persons experiencing suicidality and their families | One and a half hours
  In-depth interviews with older persons experiencing suicidality and their families - in order to understand them.

CONTACTS AND LOCATIONS:
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Israel